CLINICAL TRIAL: NCT01788280
Title: Preliminary Assessment of [18F] Fluciclatide (GE [18F]AH111585) in Glioblastoma Multiforme Treated With Bevacizumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to get materials from GE, study not proceeding and never opened to accrual
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI60947
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — Magnetic Resonance Spectroscopy; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All enrolled participants
  Interventions: Drug: Fluciclitite , PET imaging, and Bevacizumab

INTERVENTIONS:
Drug: Fluciclitite , PET imaging, and Bevacizumab — [18F] Fluciclatide and PET imaging in patients with glioblastoma multiforme (GBM) to be treated with Bevacizumab

SUMMARY:
This exploratory study uses [18F] Fluciclatide and Positron emission tomography (PET) imaging in patients with glioblastoma multiforme (GBM) to be treated with Bevacizumab. The primary objective of this study is to determine the association of [18F] Fluciclatide uptake, fludeoxyglucose (FDG) uptake, and tumor blood flow/perfusion determined with H215O and Magnetic resonance imaging (MRI) and correlate these variables with time to progression (TTP) in participants with GBM treated with Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older for inclusion in this research study. There is inadequate experience with the safety of [18F] Fluciclatide (GE [18F]AH111585) in children and therefore this radiopharmaceutical should not be used in patients under the age of 18.
* The patient must have a histologically proven GBM, and are scheduled to be treated with Avastin therapy.
* Patient has a tumor volume of > 2.0 cm in greatest diameter is required to assess response to therapy.
* An anatomic imaging study (MRI of the brain) must be current and have been obtained within 28 days prior to the research PET imaging studies.
* Patients must agree to have clinical and radiographic endpoints and the results of histopathologic tissue analysis and other laboratory information entered into a research database, as evidenced by signing the informed consent form.
* All patients, or their legal guardians, must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
* If patient is female, she must be postmenopausal for a minimum of one year, surgically sterile, or has been confirmed not to be pregnant by serum pregnancy test performed within 48 hours prior to research PET imaging.
* Patient must not be lactating.
* Pre-treatment laboratory tests for patients receiving [18F] Fluciclatide (GE [18F]AH111585) must be performed within 21 days prior to study entry.

  * These laboratory tests must be less than 4.0 times below or above the upper or lower limit range for the respective laboratory test for entry into the study (unless not medically or clinically relevant).
  * For those patients receiving coumadin or another anticoagulant the upper limit for prothrombin time or partial thromboplastin time must not exceed 6 times the upper limit of the normal range.
  * Urinalysis abnormalities will not preclude the patient from being enrolled and studied.
  * The laboratory testing will include liver enzymes (SGOT, SGPT, ALK Phos, GGT, LDH), bilirubin (total), amylase, albumin, serum electrolytes (sodium, potassium, chloride, HCO3, calcium, creatinine, urea nitrogen, glucose) CBC with platelets prothrombin time, partial thromboplastin time, BUN, creatinine and urinalysis (screening only).

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Adult patients who require monitored anesthesia for PET scanning.
* Patients who are too claustrophobic to undergo MRI or PET imaging.
* Patients with a calculated GFR of less than 30 ml/min will be excluded from the study. For a GFR between 30-60 ml/min the MRI will be possible (using half the usual administered dose of contrast) at the discretion of the study doctor. If the patient does not wish to undergo an MRI due to their renal function they will be excluded from the study.
* Patients known to be HIV positive. This is due to the unknown potential toxicities of Fluciclatide in HIV positive patients.
* Patients who cannot undergo MRI imaging due to MRI exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 36 months
  The first exploratory hypothesis to be tested is that increased [18F] Fluciclatide uptake at baseline imaging may be correlated with a shorter time to progression.

SECONDARY OUTCOMES:
Change in standardized uptake value (SUV) | 36 months
  A second exploratory hypothesis to be tested is that a larger change in [18F] Fluciclatide uptake (change in SUV) after treatment with Bevacizumab for various lengths of time is correlated with a longer time to progression. In addition more pronounced changes in FDG uptake, blood flow, and MR perfusion parameters may also correlate with a longer time to progression.

CONTACTS AND LOCATIONS:
Overall Officials: John Hoffman, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States